CLINICAL TRIAL: NCT00741390
Title: Evaluation of Blood Volume and Perceived Pain During Fingerstick Monitoring of Blood Glucose When Using Different Currently Marketed Lancing Devices and Lancets
Brief Title: Evaluation of Blood Volume and Perceived Pain During Fingerstick Monitoring of Blood Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Kenneth Kassler-Taub. MD, BD, Diabetes Care
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: BDDC-08-001
Record Dates: First submitted 2008-08-22; First posted 2008-08-26 (Estimated); Results first posted 2010-03-10 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-03

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: Diabetes; Lancets; Pain
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm A (Other): In Visit 1 subjects tested BD/33G, OTM/33G, and OTM/28G devices. In Visit 2 subjects tested BD/33G and OTM/28G. See purpose for additional information.
  Interventions: Device: BD/33G; Device: OTM / 33G; Device: OTM/28G
- Arm B (Other): In Visit 1 subjects tested BD/33G, OTM/33G and OTU/28G devices. In Visit 2 subjects tested BD/33G and OTU/28G. See purpose for additional information.
  Interventions: Device: BD/33G; Device: OTM / 33G; Device: OTU/28G
- Arm C (Other): In Visit 1 subjects tested BD/33G, OTM/33G and ACC/28G devices. In Visit 2 subjects tested BD/33G and ACC/28G. See purpose for additional information.
  Interventions: Device: BD/33G; Device: OTM / 33G; Device: ACC/28G
- Arm D (Other): In Visit 1 subjects tested BD/33G, OTM/33G and OTM/28G devices. In Visit 2 subjects tested OTM/33G and OTM/28G. See purpose for additional information.
  Interventions: Device: BD/33G; Device: OTM / 33G; Device: OTM/28G

INTERVENTIONS:
Device: BD/33G — BD Lancet device/BD 33G lancets (BGM measured with the OneTouch® UltraMini™ (BGM) and OneTouch® Ultra® test strips)
Device: OTM / 33G — OneTouch® Mini Lancet device / BD 33G lancet (BGM measured with the OneTouch® UltraMini™ (BGM) and OneTouch® Ultra® test strips)
Device: OTU/28G — OneTouch® UltraSoft® Lancet device/OneTouch® UltraSoft® 28G Lancet (BGM measured with the OneTouch® UltraMini™ BGM) and OneTouch® Ultra® test strips)
  Arms: Arm B
Device: ACC/28G — Accu-Chek® Softclix Lancet device/Accu-Chek® Softclix 28G Lancet (BGM measured with Accu-Chek® Advantage BGM and Accu-Chek® Comfort Curve test strip)
  Arms: Arm C
Device: OTM/28G — OneTouch® Mini Lancet device / OneTouch® UltraSoft® 28G Lancet (BGM measured with the OneTouch® UltraMini™ (BGM) and OneTouch® Ultra® test strips)
  Arms: Arm A; Arm D

SUMMARY:
The procurement of blood for SMBG, usually via a finger stick, is considered by many patients to be the most painful portion of diabetes therapy. This has led to the marketing of smaller gauge lancets, lancing devices with variable depth settings and blood glucose sensors that require less blood for measurement.

In this study, two main outcomes were evaluated: The first, which was assessed at Visit 1, was whether specific combinations of lancets and lancing devices would yield sufficient blood volume to allow valid assessment of diabetic subjects' glucose levels. The other outcome, assessed at Visit 2, was the level of pain perceived by subjects during lancing with specific combinations of lancets and lancing devices. During Visit 2, pain assessment was done using a Visual Analog Scale and such that for each lancet/lancing device, the lowest lancing device setting that yielded a valid BG reading for each subject during Visit 1 was used. A third outcome measure, overall comfort with lancing, was also assessed at Visit 2.

A total of 5 combinations of lancets and lancing devices were evaluated.

These were as follows:

* BD/33G = BD Lancet device/BD 33G lancets (BGM measured with the OneTouch® UltraMini™ (BGM) and OneTouch® Ultra® test strips)
* OTM/33G =OneTouch® Mini Lancet device / BD 33G lancet (BGM measured with the OneTouch® UltraMini™ (BGM) and OneTouch® Ultra® test strips)
* OTM/28G =OneTouch® Mini Lancet device / OneTouch® UltraSoft® 28G Lancet (BGM measured with the OneTouch® UltraMini™ (BGM) and OneTouch® Ultra® test strips)
* OTU/28G = OneTouch® UltraSoft® Lancet device/OneTouch® UltraSoft® 28G Lancet (BGM measured with the OneTouch® UltraMini™ (BGM) and OneTouch® Ultra® test strips)
* ACC/28G= Accu-Chek® Softclix Lancet device/Accu-Chek® Softclix 28G Lancet (BGM measured with Accu-Chek® Advantage BGM and Accu-Chek® Comfort Curve test strip)

After enrollment and qualification, subjects were assigned to one of 4 intervention arms. The arm assignment determined which 3 of the 5 combinations of lancets and lancing devices the subjects would evaluate in Visit 1 (for volume adequacy) and of these 3, which 2 they would evaluate in Visit 2 (pain during lancing). The lancet/lancing device combinations assigned to each arm are shown in the Assigned Interventions Table below.

ELIGIBILITY:
Inclusion Criteria:

* Must currently be diagnosed with either Type I or Type II diabetes mellitus.
* Must currently be performing self monitoring of blood glucose
* Must be between 18-70 years of age (inclusive).
* Must be able to read and follow study instructions in English.

Exclusion Criteria:

* Pregnant (self reported)
* History of poor blood circulation.
* Any skin condition on his or her fingers that prevents blood sampling.
* History of a bleeding disorder.
* Neuropathy or other condition affecting sensation in the hands.
* Self-reported blood borne infection (e.g., HIV, hepatitis B or C [non A, non B], syphilis, malaria, babesiosis, brucellosis, leptospirosis, arboviral infections, relapsing fever, T lymphotropic virus Type 1, Creutzfeldt-Jakob disease).
* Currently participating in another study
* Employed by BD, J&J, Roche or the Clinical Site.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2008-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Casser, MD, Principal Investigator — TKL Research, Inc.; Ronald L Rizer, PhD, Principal Investigator — Thomas J. Stephens & Associates
Locations (4):
- United States (4):
  - Thomas J. Stephens & Associates, Colorado Springs, Colorado
  - TKL Research, Inc., Carlstadt, New Jersey
  - TKL Research, Inc, Paramus, New Jersey
  - TKL Research, Inc., Ramsey, New Jersey

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 250 subjects were enrolled in this study between 8/4/2008 (first subject visit) and 9/5/2008 (last subject visit) at two study centers.
Pre-assignment Details: After enrollment, baseline characteristics such as demography, diabetes history, and current lancets were recorded for each subject. No additional baseline measures were taken. Thereafter, subjects were assigned to one of the 4 intervention arms. Subjects were able to complete the enrollment visit and Study Visit 1 activities on the first day.
Groups:
- Arm A: Visit1 (V1) Device: BD/33G,OTM/33G,OTM/28G; Visit2 (V2) Device: BD/33G,OTM/28G. The arm assignment determined which 3 of the 5 combinations of lancets and lancing devices the subjects would evaluate in Visit 1 (for volume adequacy) and of these 3, which 2 they would evaluate in Visit 2 (pain during lancing). The lancet/lancing device combinations assigned to Arm A are: Device 1: BD/33G (BD Lancet device/BD 33G lancets (BGM measured with the OneTouch® UltraMini™ (BGM) and OneTouch® Ultra® test strips) Device 2: OTM/33G (OneTouch® Mini Lancet device / BD 33G lancet (BGM measured with the OneTouch® UltraMini™ (BGM) and OneTouch® Ultra® test strips) Device 3: OTM/28G (OneTouch® Mini Lancet device / OneTouch® UltraSoft® 28G Lancet (BGM measured with the OneTouch® UltraMini™ (BGM) and OneTouch® Ultra® test strips. For Visit 2 only the BD/33G and OTM/28G were used.
- Arm B: Visit 1 (V1):BD/33G,OTM/33G,OTU/28G; Visit 2 (V2):BD/33G, OTU/28G The arm assignment determined which 3 of the 5 combinations of lancets and lancing devices the subjects would evaluate in Visit 1 (for volume adequacy) and of these 3, which 2 they would evaluate in Visit 2 (pain during lancing).The lancet/lancing device combinations assigned to Arm B are: Device 1: BD/33G (BD Lancet device/BD 33G lancets (BGM measured with the OneTouch® UltraMini™ (BGM) and OneTouch® Ultra® test strips) Device 2: OTM/33G (OneTouch® Mini Lancet device / BD 33G lancet (BGM measured with the OneTouch® UltraMini™ (BGM) and OneTouch® Ultra® test strips) Device 3: OTU/28G (OneTouch® UltraSoft® Lancet device/OneTouch® UltraSoft® 28G Lancet (BGM measured with the OneTouch® UltraMini™ (BGM) and OneTouch® Ultra® test strips). For Visit 2 only the BD/33G and OTU/28G were used.
- Arm C: Visit 1 (V1): BD/33G, OTM/33G,ACC/28G Visit 2 (V2): BD/33G, ACC/28G The arm assignment determined which 3 of the 5 combinations of lancets and lancing devices the subjects would evaluate in Visit 1 (for volume adequacy) and of these 3, which 2 they would evaluate in Visit 2 (pain during lancing). The lancet/lancing device combinations assigned to Arm C are: Device 1: BD/33G (BD Lancet device/BD 33G lancets (BGM measured with the OneTouch® UltraMini™ (BGM) and OneTouch® Ultra® test strips) Device 2: OTM/33G (OneTouch® Mini Lancet device / BD 33G lancet (BGM measured with the OneTouch® UltraMini™ (BGM) and OneTouch® Ultra® test strips) Device 3: ACC/28G (Accu-Chek® Softclix Lancet device/Accu-Chek® Softclix 28G Lancet (BGM measured with Accu-Chek® Advantage BGM and Accu-Chek® Comfort Curve test strip). For Visit 2 only the BD/33G and ACC/28G were used.
- Arm D: Visit1 (V1): BD/33G,OTM/33G,OTM/28G; V2: OTM/33G, OTM/28G The arm assignment determined which 3 of the 5 combinations of lancets and lancing devices the subjects would evaluate in Visit 1 (for volume adequacy) and of these 3, which 2 they would evaluate in Visit 2 (pain during lancing). The lancet/lancing device combinations assigned to Arm D are: Device 1: BD/33G (BD Lancet device/BD 33G lancets (BGM measured with the OneTouch® UltraMini™ (BGM) and OneTouch® Ultra® test strips) Device 2: OTM/33G (OneTouch® Mini Lancet device / BD 33G lancet (BGM measured with the OneTouch® UltraMini™ (BGM) and OneTouch® Ultra® test strips) Device 3: OTM/28G (OneTouch® Mini Lancet device / OneTouch® UltraSoft® 28G Lancet (BGM measured with the OneTouch® UltraMini™ (BGM) and OneTouch® Ultra® test strips). For Visit 2 only the OTM/33G and OTM/28G were used.
Period: Visit 1
Arm/Group | Arm A | Arm B | Arm C | Arm D
Started | 62 | 63 | 62 | 63
Completed | 60 | 63 | 55 | 62
Not Completed | 2 | 0 | 7 | 1
Period: Visit 2
Arm/Group | Arm A | Arm B | Arm C | Arm D
Started | 59 (1 subject lost to follow-up between Visit 1 and Visit 2.) | 61 (2 subjects lost to follow-up between Visit 1 and Visit 2.) | 55 | 61 (1 subject lost to follow-up between Visit 1 and Visit 2.)
Completed | 59 | 61 | 54 | 60
Not Completed | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Arm/Group | Entire Study Population
Number analyzed (Participants) | 250
Age Continuous [Mean (Standard Deviation); unit: years] | 52.1 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151
  Male | 99
Region of Enrollment [Number; unit: participants]
  United States | 250
Blood Glucose Meter Brand [Number; unit: participants]
  Abbott | 45
  Agamatrix | 1
  BD/Novamax | 17
  Bayer | 20
  Lifescan | 106
  Private Label Walgreens | 2
  Reli-on | 2
  Roche | 41
  Other | 16
Diabetes Type [Number; unit: participants]
  Type 1 | 95
  Type 2 | 155
Years Since Diagnosis [Number; unit: participants]
  <1 | 12
  1-5 | 46
  6-10 | 46
  >10 | 146

OUTCOME MEASURES:

1. Primary Outcome: Blood Sample of Sufficient Volume to Yield a Valid Meter Reading
Description: Number of subjects in whom valid meter reading was obtained with each device configuration. The primary outcome of a successful lancing is defined as whether or not a technician is able to use the lancing system to yield a blood sample of sufficient volume to yield a valid meter reading.
Time Frame: Study Day 1 (Visit 1)
Population: BD/BD33g and Mini/BD33g were included in 4 arms,the Mini/OT28g in 2 arms,and Ultra/OT28g and AC/AC28g in 1 arm. Thus the # of subj evaluated for each device was 246, 246, 124, 63, and 60, resp. Subj were analyzed for blood volume adequacy if they completed the depth setting/volume testing for at least 1 device w/o significant protocol deviation.
Measure: Number; unit: Participants
Groups:
- BD/33G: BD Lancet Device / BD 33 Gauge Lancet.
  In Study Visit 1 each subject was randomly assigned to one of four groups, each subject evaluated three different lancet device/lancet combinations. The order of evaluation of the three systems was randomly assigned for each subject. Subjects started at the middle depth setting of each lancet device. The lowest depth setting for each system yielding sufficient volume for each system was recorded for that subject and used during Visit 2. All subjects whom obtained adequate sample volumes were selected to participate in Study Visit 2.
- OTM/33G: OneTouch Mini Device / BD 33 Gauge Lancet
  See description for BD/33G.
- OTM/28G: OneTouch Mini Device / OneTouch UltraSoft 28G Lancet
  See description for BD/33G.
- OTU/28G: OneTouch UltraSoft Device / OneTouch UltraSoft 28G Lancet
  See description for BD/33G.
- ACC/28G: Accu-Chek Softclix Device / Accu-Chek Softclix 28G Lancet
  See description for BD/33G.
Arm/Group | BD/33G | OTM/33G | OTM/28G | OTU/28G | ACC/28G
Number analyzed (Participants) | 246 | 246 | 124 | 63 | 60
Participants
  Sufficient Volume - Success | 245 | 246 | 124 | 63 | 60
  Sufficient Volume - Unsuccessful | 1 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: BD/33G; Test type: Superiority or Other; Percentage = 99.59, 95% CI [98.09 to 99.59]
Statistical Analysis 2: Comparison: OTM/33G; Test type: Superiority or Other; Percentage = 100, 95% CI [98.79 to 100]
Statistical Analysis 3: Comparison: OTM/28G; Test type: Superiority or Other; Percentage = 100, 95% CI [97.61 to 100]
Statistical Analysis 4: Comparison: OTU/28G; Test type: Superiority or Other; Percentage = 100, 95% CI [95.36 to 100]
Statistical Analysis 5: Comparison: ACC/28G; Test type: Superiority or Other; Percentage = 100, 95% CI [95.13 to 100]

2. Primary Outcome: Difference in Lancing Pain for Device Pair at Visit 2. (For Subjects Assigned to Arms A, B, C Only)
Description: In Visit 2 subjects kept the same group assignment they had in Visit 1. Each subject tested 2 of the 3 systems from Visit 1. Up to 6 pairs of lancings were performed in order to obtain 4 evaluable pairs. After each pair of lancing, the subject was asked to record the pain from the 2nd lancing as compared to the first using a 150mm visual analog scale(0mm = same pain, -75mm = max score for less painful than first lancing,+75mm = max score for more painful). A positive value on the scale (and in table below) indicates that the first device in the pair was more painful than the second.
Time Frame: Approximately Day 3 (Visit 2)
Population: Of the 234 subjects that completed Visit 2, 229 had evaluable pairs and were included in the analysis for Visit 2. Some of the lancing pairs from several subjects were excluded due to protocol deviations, subject discontinuation or adverse events. Of these 175 subjects were analyzed for this primary outcome.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- OTM/28G - BD/33G: OneTouch Mini Device/OneTouch UltraSoft 28G Lancet as compared to BD Lancet Device / BD 33G Lancet
- OTU/28G - BD/33G: OneTouch UltraSoft Device/OneTouch UltraSoft 28G Lancet as compared to BD Lancet Device / BD 33G Lancet
- ACC/28G - BD/33G: Accu-Chek Softclix Device/Accu-Chek Softclix 28G Lancet as compared to BD Lancet Device / BD 33G Lancet
Arm/Group | OTM/28G - BD/33G | OTU/28G - BD/33G | ACC/28G - BD/33G
Number analyzed (Participants) | 59 | 61 | 55
mm | 10.86 (34.07) | 8.71 (36.69) | -0.03 (31.83)
Statistical Analysis 1: Comparison: OTM/28G - BD/33G; Test type: Superiority or Other; p < 0.001, ANOVA; A general linear model with subject as a random effect and order within a pair as a fixed effect was fit to each study group; Mean Difference (Net) = 10.84, 95% CI [6.80 to 10.84]
Statistical Analysis 2: Comparison: OTU/28G - BD/33G; Test type: Superiority or Other; p = 0.003, ANOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 8.55, 95% CI [3.63 to 8.55]
Statistical Analysis 3: Comparison: ACC/28G - BD/33G; Test type: Superiority or Other; p = 0.460, ANOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 0.23, 95% CI [-3.57 to 0.23]

3. Secondary Outcome: Difference in Lancing Pain for Devices in Visit 2 Only. (For Subjects Assigned to Arm D Only)
Description: The subjects who participated in Study Visit 2 kept the same group assignment they had in Study Visit 1. Each subject tested 2 of the 3 systems they experienced during Visit 1. Up to 6 pairs of lancings were performed in order to obtain 4 evaluable pairs.
  After each pair of lancing, the subject was asked to record the difference in the pain they perceive between two lancing systems using the 150 mm visual analog scale. A positive value on the scale (and in the table below) indicates that the first device in the pair was more painful than the second.
Time Frame: Approximately Day 3 (Visit 2)
Population: 61 subjects in this arm completed visit 1 and evaluable data for lancing pain. See further description above.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- OTM/28G - OTM/33G: OneTouch Mini Device/OneTouch UltraSoft 28G Lancet as compared to OneTouch Mini Device / BD 33G Lancet
Arm/Group | OTM/28G - OTM/33G
Number analyzed (Participants) | 61
mm | 4.86 (33.75)
Statistical Analysis 1: Comparison: OTM/28G - OTM/33G; Test type: Superiority or Other; p = 0.017, ANOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 4.90, 95% CI [1.14 to 4.90]

4. Secondary Outcome: Reported Device Preference Within Lancing Pair at Visit 2
Description: After each pair of 4 lancings, the subject was asked: "Which of the two devices did you find more comfortable, overall?" The choices were: first lancing, second lancing or equivalent. The "Stated Preference" row indicates # of lancing pairs in which one device was preferred over the other device while the 2 rows below indicate the # of pairs in which each device was preferred. First and second device refers to the 1st and 2nd devices identified in column headers, not the device order during testing. The "No Preference" row includes lancing pairs with preference of "equivalent" or no answer.
Time Frame: Approximately Day 3 (Visit 2)
Population: Comfort was analyzed per lancing pairs. 236 subjects performed up to 4 lancing pairs. 869 pairs were evaluated across the 4 arms. Pairs were excluded if they did not result in a valid meter reading or associated with protocol deviations or had missing comfort data.
Measure: Number; unit: lancing pairs
Groups:
- OTM/28G - BD/33G: OneTouch Mini Device / OneTouch UltraSoft 28G Lancet - BD Lancet Device / BD 33 gauge Lancet
- OTU/28G - BD/33G: OneTouch UltraSoft Device / OneTouch UltraSoft 28G Lancet - BD Lancet Device / BD 33 gauge Lancet
- ACC/28G - BD/33G: Accu-Chek Softclix Device / Accu-Chek Softclix 28G Lancet - BD Lancet Device / BD 33 gauge Lancet
- OTM/28G - OTM/33G: OneTouch MiniDevice / OneTouch 28g Lancet - OneTouch MiniDevice /BD 33 Gauge Lancet
Arm/Group | OTM/28G - BD/33G | OTU/28G - BD/33G | ACC/28G - BD/33G | OTM/28G - OTM/33G
Number analyzed (Participants) | 59 | 61 | 55 | 61
lancing pairs
  # of pairs in which participants stated preference | 180 | 183 | 173 | 186
  First device in pair preferred | 67 | 70 | 84 | 73
  Second device in pair preferred | 113 | 113 | 89 | 113
  # of pairs in which no preference was stated | 43 | 26 | 32 | 46
Statistical Analysis 1: Comparison: OTM/28G - BD/33G; Analysis consisted of a one proportion test for the 1st device in the lancing pair being preferred, out of the total number of times that a preference was stated. Note: lancing pairs in which no preference was stated or where data were missing were excluded from analysis. The null hypothesis for the one proportion test was that the 1st device in the lancing pair was preferred 50% of the times; Test type: Superiority or Other; p = 0.001, Fisher Exact; One proportion two-sided test; p=50%
Statistical Analysis 2: Comparison: OTU/28G - BD/33G; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.002, Fisher Exact; One proportion two-sided test; p=50%
Statistical Analysis 3: Comparison: ACC/28G - BD/33G; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.761, Fisher Exact; One proportion two-sided test; p=50%
Statistical Analysis 4: Comparison: OTM/28G - OTM/33G; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.004, Fisher Exact; One proportion two-sided test; p=50%

ADVERSE EVENTS:
Time Frame: Up to 1 month. At each study contact, subjects were questioned in an open-ended manner regarding any new or worsening undesirable effects that may have occurred since the previous contact. All findings were documented and evaluated by the PI or designee.
Groups:
- Arm A: Visit1 (V1) Device: BD/33G,OTM/33G,OTM/28G; Visit2 (V2) Device: BD/33G,OTM/28G
- Arm B: Visit 1 (V1) Device: BD/33G,OTM/33G,OTU/28G; Visit 2 (V2) Device: BD/33G,OTU/28G
- Arm C: Visit 1 (V1) Device: BD/33G,OTM/33G,ACC/28G; Visit 2 (V2)-BD/33G,ACC/28G
- Arm D: Visit 1 (V1) Device: BD/33G,OTM/33G,OTM/28G; Visit (V2) Device: OTM/33G,OTM/28G
Arm/Group | Arm A | Arm B | Arm C | Arm D
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/63 | 0/62 | 0/63
Other Adverse Events (participants affected / at risk) | 5/62 | 6/63 | 11/62 | 6/63
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=62) | Arm B (N=63) | Arm C (N=62) | Arm D (N=63)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 7 (7) | 2 (2)
hypoglycemia (Metabolism and nutrition disorders) | 4 (6) | 5 (6) | 4 (5) | 4 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less